CLINICAL TRIAL: NCT04637893
Title: The Impact of Covid-19 Pandemic on Colorectal Cancer Prevention Due to Delays in Diagnosis: a Global Study
Acronym: COVID_CRC
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 100
Record Dates: First submitted 2020-11-18; First posted 2020-11-20 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Colonoscopy — Pt. underwent colonoscopy

SUMMARY:
Screening programs have been associated with a substantial reduction in colorectal cancer (CRC) mortality through endoscopic resection of preneoplastic lesions and detection of early-stage invasive cancers.

In March 2020, the World Health Organization declared as a pandemic the outbreak of coronavirus disease 2019 (COVID-19), caused by SARS-CoV-2. Since then, the SARS-CoV-2 have never stopped spreading, causing an unprecedented situation with highly restrictive considerations to be adopted by the majority of countries worldwide.

Health-care facilities have been making an enormous effort to assist patients affected by COVID-19, while adopting measures to maintain a safe environment for patients and healthcare professionals. As a result, the usual workflow in endoscopy departments changed dramatically, leading to an increase in cancelled procedures, probably increasing the future burden of Colorectal Cancer due to delays in diagnosis.

ELIGIBILITY:
* patients who underwent colonoscopy between the 1st October 2020 and the 31st December 2020 (pandemic cohort)
* patients who underwent colonoscopy between the 1st October 2019 and the 31st December 2019 (pre-pandemic cohort)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent colonoscopy between the 1st October 2020 and the 31st December 2020 (pandemic cohort), and all patients who underwent colonoscopy between the 1st October 2019 and the 31st December 2019 (pre-pandemic cohort).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Colorectal Cancer prevention | 3 months
  To investigate the impact of COVID-19 pandemic on Colorectal Cancer prevention on a global scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — IRCSS Humanitas Research Hospital
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No